CLINICAL TRIAL: NCT00118768
Title: A Randomized, Phase IIb Clinical Trial to Evaluate the Safety and Antiviral Activity of the Combination of Pegylated Interferon Alfa Plus NM283 (Valopicitabine) in Treatment-Naive Patients With Chronic Hepatitis C
Brief Title: A Study to Evaluate the Combination of Pegylated Interferon Alfa Plus Valopicitabine in Patients With Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-08A-006
Record Dates: First submitted 2005-06-30; First posted 2005-07-12 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype-1, Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — valopicitabine

INTERVENTIONS:
Drug: valopicitabine
Drug: Pegylated Interferon Alfa

SUMMARY:
This Phase II study is being conducted in treatment-naive patients (no previous antiviral therapy for Hepatitis C infection) with genotype-1 chronic hepatitis C to evaluate the safety and effectiveness of valopicitabine alone and together with Pegylated Interferon (a drug approved by the Food and Drug Administration for the treatment of Hepatitis C infection).

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history of genotype-1 chronic Hepatitis C and compensated liver disease
* Treatment Naive (patient has received no previous treatment for chronic hepatitis C infection)
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with HIV or Hepatitis B
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Phoenix, Arizona
  - San Diego, California
  - San Mateo, California
  - Lakewood, Colorado
  - Bradenton, Florida
  - Gainesville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Laurel, Maryland
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Kansas City, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
  - San Antonio, Texas
  - Tacoma, Washington